CLINICAL TRIAL: NCT04053491
Title: Comparison of the Infraclavicular and Axillary Approaches for Continuous Ultrasound-guided Brachial Plexus Block: A Prospective Randomized Study
Brief Title: Comparison of the Infraclavicular and Axillary Approaches for Continuous Ultrasound-guided Brachial Plexus Block.
Acronym: ICAX
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: funding not obtained
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUBX 2019/04
Record Dates: First submitted 2019-08-07; First posted 2019-08-12 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Anesthesia, Regional; Brachial Plexus Block
Keywords: Hand surgery; Anesthesia, Regional; Brachial Plexus Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Axillary block group (Experimental): Initial bolus will be given and then a perinervous catheter will be inserted by the axillary approach.
  Interventions: Procedure: Hand surgery under regional anesthesia
- Infraclavicular block group (Experimental): Initial bolus will be given and then a perinervous catheter will be inserted by the infraclavicular approach.
  Interventions: Procedure: Hand surgery under regional anesthesia

INTERVENTIONS:
Procedure: Hand surgery under regional anesthesia — In both groups, patients will benefit from an initial standardized bolus (long-acting local anesthetic, ropivacaine) to cover the operative period, via the allocated approach. Ultrasound guidance and the recommended standards monitors will be used in both groups. After the initial bolus, a catheter will be inserted via the allocated approach. Surgery will be done under regional anesthesia alone, unless there is a medical contraindication or if the patient asks for general anesthesia. Post-operative analgesia will be standardized with regular paracetamol, regular NSAID (Nonsteroidal anti-inflammatory drugs) and oxycodone if needed. The local anesthetics perfusion will be standardized. There will be a medical follow up at 24 and 48 hours where data will be collected.

SUMMARY:
Prospective randomized study comparing the axillary and the infraclavicular approaches for continuous brachial plexus block after hand surgery.

DETAILED DESCRIPTION:
Regional anesthesia is considered as the gold standard for analgesia and anesthesia of hand surgeries. However, with a single-shot technique, a maximum of 13 hours of analgesia is obtained, even with a long-acting local anesthetic and adjuvants. For painful surgeries necessitating prolonged analgesia of more than 24 hours, continuous regional analgesia techniques have been described, using perinervous catheters. However, these techniques have a high incidence of failure. The most frequent causes of failure are catheter displacements, misplacement, and the distance between the targeted nerves. Many approaches have been described to insert these catheters (axillary, infraclavicular and supraclavicular), but the optimal approach remains unknown. Therefore, international and even local practices vary widely.

Investigators plan to compare the axillary and the infraclavicular approaches in this randomized study, on 60 patients. In every group, an initial bolus will be given and then a perinervous catheter will be inserted by the allocated approach. The surgery will be done under regional anesthesia. The co-analgesia, the local anesthetic infusion and the follow-up will be standardized and will be the same in the two groups.

The primary outcome will be an anesthesia score on 16 points previously described in other similar publication. The primary outcome will be at 24 hours after block realization, but it will be repeated at 48 hours. It will evaluate the degree of sensitive and motor blockade of every major nerve of the hand. Secondary outcomes will be the time, comfort and adverse effects of the technique, and postoperative pain, analgesia, satisfaction and adverse effects.

The aim of this study is to help determine the optimal approach for brachial plexus catheter insertion, in order to improve analgesia, to decrease morphine consumption and its related adverse effects, and to improve patients and caregivers satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a social insurance number
* ASA 1-3
* Patients undergoing hand surgery requiring a continuous brachial plexus block
* Elective or urgent surgery
* Effective contraception (HAS criteria)
* Informed consent

Exclusion Criteria:

* Contraindication to the installation of a continuous brachial plexus block (coagulopathy, refusal, allergy to the medication)
* Preexisting neuropathy
* Pregnancy
* Arteriovenous fistula
* Obesity (BMI >40)
* Another surgical site implicated during the surgery
* Incapacity to abduct the operated arm
* Preoperative use of morphine or equivalent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Anesthesia score | 24 hours after block realization
  Min/Max : 0 for no anesthesia to 16 total anesthesia Addition of Motor block score (0-2) and Sensitive block score (0-2) for the 4 main nerves of the hand

SECONDARY OUTCOMES:
Duration of catheter insertion procedure | During block realization
Maximal pain during the surgery procedure | During surgery
  Measured by patient with numeric scale from 0 = no pain to 10 = maximal pain
Maximal pain during the first 24 hours | During the first 24 hours after block realization
  Measured by patient with numeric scale from 0 = no pain to 10 = maximal pain
Anesthesia score | 30 minutes after block realization
  Min/Max : 0 for no anesthesia to 16 total anesthesia Addition of Motor block score (0-2) and Sensitive block score (0-2) for the 4 main nerves of the hand
Anesthesia score | 48 hours after block realization
  Min/Max : 0 for no anesthesia to 16 total anesthesia Addition of Motor block score (0-2) and Sensitive block score (0-2) for the 4 main nerves of the hand
Total morphine consumption | 24 and 48 hours after block realization
Mean pain at rest and with movement | 24 and 48 hours after block realization
  Measured by patient with numeric scale from 0 = no pain to 10 = maximal pain
Quality of sleep | Over first night after block realization
  Measured by patient with numeric scale from 0 = insomnia to 10 = excellent sleep
Patient satisfaction | 48 hours after block realization
  Measured by patient with numeric scale from 0 = fully unsatisfied to 10 = fully satisfied

IPD SHARING:
Plan to Share IPD: No